CLINICAL TRIAL: NCT03931590
Title: Phase 1 Study to Investigate the Absorption, Metabolism, and Excretion of [14C] Omaveloxolone Following Single Oral Dose Administration in Healthy Male Subjects
Brief Title: A Human AME Study for Omaveloxolone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 408-C-1805
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Healthy Male Subjects
Keywords: RTA 408; RTA 408 capsules; omaveloxolone; omaveloxolone capsules; AME; mass balance; metabolite identification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Healthy Male Subjects (Experimental): Single oral dose of 150 mg of [14C] omaveloxolone containing approximately 90 μCi as a capsule after an overnight fast of at least 10 hours.
  Interventions: Drug: [14C]-Omaveloxolone

INTERVENTIONS:
Drug: [14C]-Omaveloxolone — [14C]-Omaveloxolone 50 mg capsules
  Other Names: [14C]-RTA 408

SUMMARY:
This study will assess the pharmacokinetics (PK), mass balance, metabolite profiles, and rates and routes of elimination of [14C] omaveloxolone and derived metabolites following administration as a single 150 mg (containing approximately 90 µCi) dose to healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy all of the following criteria at the Screening Visit unless otherwise stated:
* Males, of any race, between 18 and 55 years of age, inclusive.
* Body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive, and a total body weight > 50 kg.
* Be surgically sterile or willing to agree to use contraception
* In good health, as assessed by the investigator (or designee).
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Exclusion Criteria:

* Significant history or clinical manifestation of any major system disorder, as determined by the investigator (or designee).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs.
* Presence of any other condition, including surgery, known to interfere with the absorption, distribution, metabolism, or excretion of medicines.
* Abnormal laboratory values considered clinically significant by the investigator.
* Clinically significant abnormal 12-lead ECGs.
* History of alcoholism or drug/chemical abuse within 2 years prior to Check-in (Day-1).
* Alcohol consumption of > 21 units per week.
* Positive urine drug screen at Screening, or positive alcohol breath test result or positive urine drug screen at Check-in (Day -1).
* Positive hepatitis panel and/or positive human immunodeficiency virus test.
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives (if known) prior to dosing.
* Current enrollment in another clinical study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of omaveloxolone | 22 days
  Pharmacokinetics will be assessed by blood sampling for omaveloxolone to determine maximum observed concentration (Cmax).
Area under the omaveloxolone concentration-time curve (AUC) | 22 days
  Pharmacokinetics will be assessed by blood sampling for omaveloxolone to determine area under the curve (AUC).
Maximum concentration of total radioactivity in blood and plasma | 22 days
  Mass balance and metabolite profiles will be assessed by blood sampling for omaveloxolone to determine maximum concentration of total radioactivity
Area under the concentration-time curve total radioactivity in blood and plasma | 22 days
  Mass balance and metabolite profiles will be assessed by blood sampling for total radioactivity to determine area under the concentration-time curve.
Amount of radioactivity excreted in urine (Aeu) | 22 days
  Rates and routes of elimination will be assessed by urine sampling for radioactivity.
Amount of radioactivity excreted in feces (Aef) | 22 days
  Rates and routes of elimination will be assessed by sampling of feces for radioactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Siebers, MD, Principal Investigator — Covance CRU Inc.
Locations (1):
- Covance Clinical Research Unit (CRU) Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/